CLINICAL TRIAL: NCT05175183
Title: Epidemiology of Speed Skating-related Injuries
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, PhD, University of Oviedo
Other Study IDs: UO2021-04
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Sports Injury
Keywords: Prevalence; Multidirectional Sport; Injury prevention; Athletic injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Speed skating is a sport in which there´s a lack of epidemiological studies. In line with the well-established model of sports injury prevention research proffered by van Mechelen, the first stage in this process is establishing the extent of the problem i.e. injury incidence, severity and burden. Through an online survey filled by semiprofessional athletes, it is posible to obtain all this important information. This way, it will be possible to fulfill a gap in the literature and take action in the near future in order to reduce the prevalence of injuries in this sport.

DETAILED DESCRIPTION:
A retrospective study will be performed in speed skaters. 100 speed skaters will be recruited. Data of all injury along a whole season will be collected. Patients' information, including age, number of years playing, skill level and injured body part, will be analysed

ELIGIBILITY:
Inclusion Criteria:

* Being a speed skater and having competed in the 2018 spanish national championship

Exclusion Criteria:

* Being unable to understand the questionaire, do not accept on participating in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Speed skaters competing in the spanish national championship
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
1.Injury prevalence | [Time Frame: January 2018-December 2018]
  Injury prevalence rates [Injury prevalence rates calculated per 1000 hours of play]

SECONDARY OUTCOMES:
Injury burden | [Time Frame: January 2018-December 2018]
  Days lost per 1000 hours of exposure
Injury prevalence according to occurrence | [Time Frame: January 2018-December 2018]
  Number of injuries sustained during training/ Number of injuries sustained during a match (% of all)
Injury prevalence by mechanism of injury | [Time Frame: January 2018-December 2018]
  Number of injuries according to the mechanism of injury (Contact (Direct or indirect) or Non-Contact) (% of all)
Injury prevalence according to location | [Time Frame: January 2018-December 2018]
  Distribution of injuries according to location of the injury (on the body, % of all)
Injury prevalence according to tissue affected | [Time Frame: January 2018-December 2018]
  Description of the distribution of injuries according to the type of the injury (muscle only) (% of all)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Olmedillas, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Paper published, link to access — http://doi.org/10.1123/jsr.2021-0443